CLINICAL TRIAL: NCT05463653
Title: Evaluation of the Efficacy of an Early Rehabilitation Intervention, Supported by Telemedicine, Compared to the Usual Rehabilitation Intervention, in Patients With Distal Radius Fracture. Randomized Clinical Trial
Brief Title: Comparison of Rehabilitation Intervention, Supported by Telemedicine, With Standard Rehabilitation After Distal Radius Fracture.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinico Mutual de Seguridad (Other)
Responsible Party: Principal Investigator, Felipe Andrés Correa Salazar, Physical therapist, Hospital Clinico Mutual de Seguridad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2022-07-13; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Distal Radius Fracture
Keywords: Rehabilitation; Information technologies
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Two arms parallel design, randomized assignment, outcomes-assessor blind to the assignment
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is a physical therapist independent of the research team, who is blind to the treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental telemedicine (Experimental): Patient's rehabilitation and compliance with the standard exercices will be guided and monitored through an ad hoc device developed specifically for this trial.
  Interventions: Device: Experimental
- Control (Active Comparator): Patient's rehabilitation and compliance with the standard exercices will be monitored in the usual manner, at the monthly visits to the physical therapy clinic
  Interventions: Device: Experimental

INTERVENTIONS:
Device: Experimental — A digital pad developed to help, support and monitor the adherence of patients to rehabilitation excercices post surgery

SUMMARY:
This is a randomized clinical trial of two parallel arms, aiming to compare two rehabilitation interventions: an experimental intervention including telemedicine support and remote monitoring of compliance of usual indicated exercises, versus the usual protocol of indicated exercises supported by printed material (triptych) and without remote monitoring

DETAILED DESCRIPTION:
Distal radius fracture is a common pathology. The surgical indication is given by the difficulty in obtaining fracture reduction or by the instability of the fracture. The long-term functional prognosis of the wrist depends largely on patients' adherence to the prescribed indications/exercises in the immediate postoperative phase.

This is a randomized clinical trial of two parallel arms, aiming to compare two rehabilitation interventions: an experimental intervention including telemedicine support and remote monitoring of compliance of usual indicated exercises, versus the usual protocol of indicated exercises supported by printed material (triptych) and without remote monitoring.

ELIGIBILITY:
Inclusion Criteria:

* distal radial fracture (A2 to C3 type according to the Orthopaedic Trauma Association classification system)
* indication for standard rehabilitation post-surgery

Exclusion Criteria:

* immediate post-surgery complication
* multiple fractures or severe injuries
* history of bone metabolism condition
* illiterate
* non-Spanish speaking
* mental disorder
* not familiar with electronic devices

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of Patient Related Wrist Evaluation score from Day 28 at Day 56 post ranndomization | Day 56
  Patient Related Wrist Evaluation is a 15-item validated scale, range from 0 to 100, where higher scores are worse outcomes
Adherence to prescribed excercise program | Day 56
  The digital pad will objectively register adherence to exercises; the control group will self-report their compliance rates with the prescribed exercises

SECONDARY OUTCOMES:
Grip strength | Day 28; Day 56
  Grip strength measured by dynamometer
Wrist flexion and extension | Day 28; Day 56
  Wrist flexion and extension measured by goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Gamboa, Study Director — Mutual de Seguridad General Manager
Locations (1):
- Hospital Clinico Mutual de Seguridad, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No